CLINICAL TRIAL: NCT05917743
Title: Mat Pilates vs. General Exercises for Acute Nonspecific Low Back Pain: A Randomized Controlled Trial
Brief Title: Mat Pilates Versus General Exercises for Patients With Nonspecific Acute Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/00Z001
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mat Pilates (Experimental): Mat Pilates exercises targeting core strength, flexibility, and muscle control
  Interventions: Other: Mat Pilates
- General Exercises (Active Comparator)
  Interventions: Other: General Exercises

INTERVENTIONS:
Other: Mat Pilates — Duration: 50 minutes per session Repetitions: 8-12 repetitions per exercise Sets: 2-3 sets per exercise Rests: 30-60 seconds rest between sets Frequency: 3 times per week for 4 weeks Exercises: A series of Mat Pilates exercises targeting core strength, flexibility, and muscle control
  Arms: Mat Pilates
Other: General Exercises — General exercise is a structured exercise program designed to help individuals with back pain improve their fitness levels. The program comprises of a series of exercise classes that are led by a physiotherapist. The classes involve a combination of aerobic, strength, and flexibility exercises, and aim to improve overall physical fitness, reduce pain, and improve function. The program is specifically designed for individuals with back pain, and the exercises are tailored to meet the needs of each participant. The Back to Fitness Program is based on the principles of exercise prescription and is intended to be a safe and effective way to manage back pain through exercise.
  Arms: General Exercises

SUMMARY:
Aim: To compare the effectiveness of Mat Pilates with General Exercises in treating patients with nonspecific acute low back pain.

Novelty: Pilates, typically performed with specific equipment, has shown clinically significant treatment effects in people with chronic low back pain. Recent guidelines recommend patients remain active during episodes of low back pain; however, evidence regarding the type of exercise to perform is limited. Mat Pilates is a type of Pilates exercise that does not require complex equipment. Evaluating the effectiveness of two simple exercise methods (Mat Pilates and General Exercises) can help expand intervention options for patients with acute low back pain, enabling them to choose an exercise they enjoy most.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 50 years old
* Acute nonspecific low back pain with at least 3 points on the Visual Analog Scale (VAS)
* Willing and able to provide informed consent
* Able to comply with the study protocol and attend all treatment sessions and follow-up assessments

Exclusion Criteria:

* Presence of specific low back pain causes, such as lumbar radiculopathy, spinal stenosis, or spondylolisthesis
* Previous spinal surgery
* Contraindications to exercise, such as severe cardiovascular or respiratory conditions
* Currently pregnant or planning to become pregnant during the study period
* Participation in another clinical trial or receiving concurrent experimental treatment for low back pain

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity | Change from baseline to 4 weeks and 3 months
  Pain intensity will be assessed using the Visual Analog Scale (VAS) at baseline (pre-treatment), 4 weeks after randomization (post-treatment), 3 months after discharge (follow-up 1). The VAS is a continuous scale comprising a horizontal line, anchored by two verbal descriptors, one for each symptom extreme.

SECONDARY OUTCOMES:
Change in Disability | Change from baseline to 4 weeks and 3 months
  Disability will be assessed using the Roland-Morris Disability Questionnaire (RMDQ) at baseline (pre-treatment), 10 weeks after randomization (post-treatment), 3 months after discharge (follow-up 1), and 6 months after discharge (follow-up 2). The RMDQ is a 24-item self-report questionnaire measuring level of disability/function in people with low back pain. Higher scores indicate higher disability.
Change in Pain Pressure Threshold | Change from baseline to 4 weeks and 3 months
  Pain pressure threshold will be assessed using a pressure algometer at baseline (pre-treatment), 10 weeks after randomization (post-treatment), 3 months after discharge (follow-up 1), and 6 months after discharge (follow-up 2). A pressure algometer objectively evaluates pain sensitivity levels by measuring the minimum stimulus intensity perceived as painful.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The researchers of this study are committed to promoting open science and collaboration among researchers. As part of this commitment, we will share de-identified individual participant data (IPD) with other qualified researchers, upon request and in accordance with applicable regulations and ethical guidelines.
Supporting Information: SAP, ICF
Time Frame: De-identified IPD will be available for sharing with other researchers starting six months after the publication of the primary study results and will remain accessible for a period of 2 years.
Access Criteria: via mohamed.elmeligie@acu.edu.eg